CLINICAL TRIAL: NCT02687984
Title: A Multicenter, Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of RBP-7000 Using Poly (DL-lactide-co-glycolide) Polymer of Two Different Molecular Weights (Low and High Molecular Weights as Test Treatments) Compared to Intermediate Molecular Weight (Reference Treatment) Polymer in Subjects With Schizophrenia
Brief Title: PK, Safety, and Tolerability Study of RBP-7000 of Different Molecular Weight Polymer in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-15-0001
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Long-acting Risperidone; Atrigel
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RBP-7000 PLGH A (Experimental): A single subcutaneous injection of RBP-7000 containing 120 mg risperidone in the ATRIGEL® Delivery System formulated with 21 kDa PLGH polymer.
  Interventions: Drug: RBP-7000
- RBP-7000 PLGH B (Experimental): A single subcutaneous injection of RBP-7000 containing 120 mg risperidone in the ATRIGEL® Delivery System formulated with 29 kDa PLGH polymer.
  Interventions: Drug: RBP-7000
- RBP-7000 PLGH C (Active Comparator): A single subcutaneous injection of RBP-7000 containing 120 mg risperidone in the ATRIGEL® Delivery System formulated with 26 kDa PLGH polymer. This intermediate molecular weight treatment serves as the reference treatment.
  Interventions: Drug: RBP-7000

INTERVENTIONS:
Drug: RBP-7000 — A single subcutaneous injection with doses of RBP-7000 containing 120 mg risperidone and either a low, high, or intermediate molecular weight PLGH polymer.
  Other Names: Risperdal

SUMMARY:
Primary Objective: To assess the relative bioavailability of RBP-7000 formulated with 2 different molecular weights (MW) (low and high MW as test treatments) of poly (DL-lactide-co-glycolide) with a carboxylic acid end group (PLGH) polymer compared to intermediate MW PLGH polymer following single subcutaneous (SC) injection of RBP-7000 in subjects with stable schizophrenia.

Secondary Objective:

To evaluate the safety and tolerability of single SC injections of RBP-7000 using a PLGH polymer of 2 different MW (low and high MW as test treatments) compared to intermediate MW polymer in subjects with stable schizophrenia.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, single-dose, parallel-group study in subjects with clinically stable schizophrenia who are not currently taking risperidone. A total of approximately 48 subjects (16 per group) will be randomized to receive a single subcutaneous (SC) injection of RBP-7000 120 mg formulated with PLGH polymer of either 21 kilodaltons (kDa) (low MW group), 29 kDa of PLGH polymer (high MW group), or 26 kDa of PLGH polymer (intermediate MW group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia as defined by DSM-5 criteria.
* Clinically stable schizophrenia, as evidenced by the investigator evaluation, outpatient status for at least 30 days prior to screening, and confirmation of stability by a caregiver who has regular supportive contact with the subject.
* Otherwise healthy on the basis of physical examination.
* Body mass index (BMI) between 18 and 35 kg/m^2 and weight of at least 49.9 kg at screening.

Exclusion Criteria:

* Subjects taking any oral risperidone product (except the test doses of 0.25 mg of risperidone); or subjects taking any risperidone or 9-hydroxyrisperidone sustained-release or depot formulation within 120 days prior to study screening; or subjects who have received the 3-month depot formulation of 9-hydroxyrisperidone within 2 years of study screening.
* Subjects taking a clinically relevant inducer or inhibitor of cytochrome P450 (CYP) 2D6, or CYP3A4, who have not undergone proper washout (minimum of 5 half-lives of the medication) of this prohibited medication prior to Day 1.
* Medications, which in the opinion of the Investigator in conjunction with the medical monitor, may be expected to significantly interfere with metabolism or excretion of risperidone and/or 9-hydroxyrisperidone; may be associated with a significant drug interaction with risperidone; or may pose a significant risk to a subject's participation in the study.
* Any natural products or herbal preparations including all vitamins and supplements throughout the study.
* Subjects with a history of cancer unless disease-free for ≥5 years (with the exception of resected basal cell or squamous cell carcinoma of the skin).
* Subjects with any other active medical condition/disorder/disease that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug.
* Subjects that had an exacerbation of schizophrenia in the last 30 days.
* Subjects with evidence or history (in the past 6 months prior to screening) of a significant hepatic disorder that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug, including:
* Acute or chronic hepatitis, including but not limited to hepatitis B or C.
* Total bilirubin >1.5 x the upper limit of normal (ULN), or
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x ULN.
* Subjects with a history of severe renal disease, or creatinine clearance <60 mL/min
* Subjects with evidence or history of orthostatic hypotension within 6 months of screening.
* Subjects with absolute neutrophil count <1.5x 10^9/L (African and African/American <1.2x 10^9/L).
* Subjects with a history of drug-induced leucopenia.
* Subjects who have acquired immune deficiency syndrome (AIDS) or to be human immunodeficiency virus (HIV)-positive.
* Subjects with other medical conditions including, but not limited to, history of heart attack (myocardial infarction) or brain injury (traumatic injury with loss of consciousness and/or cerebrovascular accident), or clinically significant low blood pressure or arrhythmias as interpreted by the Principal Investigator or medically qualified sub-investigator.
* Subjects with congenital long QT syndrome, history of prolonged QT in the 3 months prior to screening, or a corrected QT interval (Fridericia - QTcF) >450 msec (male) or >470 msec (female) at screening (Visit 1).
* Subjects with suicidal ideation with intent or plan
* Subjects with uncontrolled depression, in the opinion of the Investigator.
* Subjects with a diagnosis of insulin-dependent diabetes, or who have a hemoglobin A1c (HbA1c) ≥8.0% at screening, or have had changes in diabetic medication regimen in the 28 days prior to signing the informed consent document.
* Subjects with prior allergic reactions, sensitivities or other known contraindications to any component of RBP-7000 (e.g., risperidone, PLGH or NMP).
* Women of childbearing potential who are pregnant or breastfeeding, seeking pregnancy, or failing to use adequate contraceptive methods during the study.
* Subjects with the presence of opioids, cocaine, amphetamines, methadone, barbiturates, benzodiazepines, methamphetamines, cannabinoids, or phencyclidine in the urine as assessed by a urine drug screen.
* Subjects with epilepsy or other seizure disorders, Parkinson's disease or dementia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Initial Burst Parameters: Cmax of risperidone | approximately 0-24 hours; Day 1 to Day 2
  Maximum observed plasma concentration
Initial Burst Parameters: AUC0-24h of risperidone | approximately 0-24 hours; Day 1 to Day 2
  Area under the plasma concentration-time curve from time 0 to 24 hours post-dose; calculated using the linear trapezoidal rule.
Secondary Peak Parameters: Cmax of risperidone | approximately 24-672 hours; Day 2 to Day 29
  Maximum observed plasma concentration
Secondary Peak Parameters: AUCD2-D29 of risperidone | approximately 24-672 hours; Day 2 to Day 29
  Area under the plasma concentration-time curve from 24 hours post-dose (Day 2) to 672 hours post-dose (Day 29); calculated using the linear trapezoidal rule.
Overall Parameters: Cmax of risperidone | Day 1 to Day 29
  Maximum observed plasma concentration
Overall Parameters: AUCD1-D29 of risperidone | Day 1 to Day 29
  Area under the plasma concentration-time curve from time 0 (Day 1) to 672 hours post-dose (Day 29); calculated using the linear trapezoidal rule.

SECONDARY OUTCOMES:
Initial Burst Parameters: Cmax of 9-hydroxyrisperidone | approximately 0-24 hours; Day 1 to Day 2
  Maximum observed plasma concentration
Initial Burst Parameters: AUC0-24h of 9-hydroxyrisperidone | approximately 0-24 hours; Day 1 to Day 2
  Area under the plasma concentration-time curve from time 0 to 24 hours post-dose; calculated using the linear trapezoidal rule.
Secondary Peak Parameters: Cmax of 9-hydroxyrisperidone | approximately 24-672 hours; Day 2 to Day 29
  Maximum observed plasma concentration
Secondary Peak Parameters: AUCD2-D29 of 9-hydroxyrisperidone | approximately 24-672 hours; Day 2 to Day 29
  Area under the plasma concentration-time curve from 24 hours post-dose (Day 2) to 672 hours post-dose (Day 29); calculated using the linear trapezoidal rule.
Overall Parameters: Cmax of 9-hydroxyrisperidone | Day 1 to Day 29
  Maximum observed plasma concentration
Overall Parameters: AUCD1-D29 of 9-hydroxyrisperidone | Day 1 to Day 29
  Area under the plasma concentration-time curve from time 0 (Day 1) to 672 hours post-dose (Day 29); calculated using the linear trapezoidal rule.
Summary of Participants with Adverse Events | Day 1 to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Indivior Inc.
Locations (2):
- United States (2):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Collaborative Neuroscience Network, Torrance, California

IPD SHARING:
Plan to Share IPD: No